CLINICAL TRIAL: NCT03597022
Title: Multiple Escalating Dose Study of BAY1093884 in Adults With Hemophilia A or B With or Without Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to thrombosis
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19580; 2017-003324-67 (EudraCT Number)
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Hemophilia A and B
Keywords: Subcutaneous; Prophylaxis; Non-Inhibitors; Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — lipoprotein-associated coagulation inhibitor; Antibodies, Monoclonal; Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- BAY1093884 100mg (Experimental): Subjects received BAY1093884 100 mg once a week until premature termination of the study
  Interventions: Drug: Befovacimab (BAY1093884)
- BAY1093884 225mg (Experimental): Subjects received BAY1093884 225 mg once a week until premature termination of the study
  Interventions: Drug: Befovacimab (BAY1093884)
- BAY1093884 400mg (Experimental): Subjects received BAY1093884 400mg once a week until premature termination of the study
  Interventions: Drug: Befovacimab (BAY1093884)

INTERVENTIONS:
Drug: Befovacimab (BAY1093884) — Once weekly doses until premature termination of the study, subcutaneous injection
  Other Names: Anti-TFPI (Tissue Factor Pathway Inhibitor) monoclonal antibody (immunoglobulin G2; IgG2)

SUMMARY:
The purpose of this study was to assess the safety and tolerability of multiple doses of a human monoclonal antibody (BAY1093884) given under the skin in subjects with hemophilia A or B. This antibody was intended to protect from bleeds by inhibiting a substance (Tissue Factor Pathway Inhibitor, TFPI) that reduces the ability of the body to form blood clots.

DETAILED DESCRIPTION:
The primary objective of the study was to assess the safety and tolerability of multiple subcutaneous injections of BAY1093884 (anti-TFPI monoclonal antibody, immunoglobulin G2, IgG2) in patients with hemophilia A or B with or without inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Male severe hemophilic patients with undetectable FVIII activity <1% or FIX activity <2%, with or without inhibitors (any titer) are eligible.
* Subjects with a past history of inhibitors (any inhibitor titer) are eligible.
* Age ≥18 years.
* Documentation of ≥4 bleeding episodes (any type or location of bleeds, treated or not) within the 6 months prior to screening.
* For subjects on prophylaxis: Willingness to interrupt ongoing prophylaxis.
* For subjects on immune tolerance induction (ITI): Willingness to interrupt ongoing ITI.

Exclusion Criteria:

* History of any other coagulation disorder (particularly disseminated intravascular coagulopathy or combined FVIII/FV deficiency) or platelet disorder.
* History of diseases related to venous thromboembolic events (e.g., pulmonary embolism, deep vein thrombosis, thrombophlebitis) or thrombotic microangiopathy.
* Risk factors for venous or arterial diseases (e.g., uncontrolled hypertension, uncontrolled diabetes).
* History of cardiac, coronary and/or arterial peripheral atherosclerotic disease
* Platelet count <100,000/μL.
* Human immunodeficiency virus (HIV) infection with a cluster of differentiation 4 (CD4+) lymphocyte count of <200/mm^3

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Fiona Stanley Hospital, Murdoch, Western Australia, Australia
- Universitätsklinikum AKH Wien, Vienna, Austria
- Bulgaria (3):
  - Medical centre Hipokrat - N EOOD, Plovdiv
  - SHATHD Spec. Hospi. for Active Treatm. of Haematol. Dis. EAD, Sofia
  - MHAT Sveta Marina EAD, Varna
- France (2):
  - Hôpital Louis Pradel - Bron, Bron
  - Hôpital Robert Debré - Reims Cedex, Reims
- Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs, Hungary
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy, Italy
- Japan (2):
  - Ogikubo Hospital, Suginami, Tokyo
  - Hiroshima University Hospital, Hiroshima
- Haematology Service, Canterbury Health Laboratories, Christchurch, New Zealand
- Eulji University Hospital, Daejeon, South Korea
- Changhua Christian Hospital, Changhua, Taiwan
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - Royal Free Hospital, London
  - Manchester Royal Infirmary, Manchester

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in 11 countries or regions between 24 July 2018 (first subject first visit) and 15 October 2019 (last subject last visit).
Pre-assignment Details: Overall, 26 participants were screened. Of them, 1 participant was screen failure and 1 participant could not start subsequent treatment on schedule; 24 participants received study treatment.
Period: Overall Study
Arm/Group | BAY1093884 100mg | BAY1093884 225mg | BAY1093884 400mg
Started | 8 | 8 | 8
Completed | 0 | 0 | 0
Not Completed | 8 | 8 | 8
Not completed — Premature termination of the study | 7 | 7 | 8
Not completed — Serious adverse event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): all subjects with at least one intake of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | BAY1093884 100mg | BAY1093884 225mg | BAY1093884 400mg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (14.5) | 43.5 (15.6) | 43.1 (5.9) | 43.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 6 | 6 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Treatment-emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence (i.e., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant in the study. Any bleeding event occurring during the study was not documented as an AE because this event was planned to be captured in the assessment of efficacy. AEs occurring after the first administration of study drug and up to and including 30 days after the last administration of study drug were defined as treatment-emergent AEs (TEAEs). Drug-related TEAEs were TEAEs that had "reasonable causal relationship" to the study treatment decided by the investigators.
Time Frame: After the first administration of study drug and up to and including 30 days after the last administration of study drug, with an average of 183 days
Population: Safety analysis set (SAF): all participants with at least one intake of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | BAY1093884 100mg | BAY1093884 225mg | BAY1093884 400mg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 1 | 4 | 5

2. Primary Outcome: Number of Participants With Serious Treatment-emergent Adverse Events
Description: A serious adverse event (SAE) was any untoward medical occurrence that at any dose was resulting in death, was lifethreatening, requires hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity. SAEs occurring after the first administration of study drug and up to and including 30 days after the last administration of study drug were defined as serious treatment-emergent AEs (TESAEs). Drug-related TESAEs were TESAEs that had "reasonable causal relationship" to the study treatment decided by the investigators.
Time Frame: as for outcome 1
Population: Safety analysis set (SAF): all participants with at least one intake of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | BAY1093884 100mg | BAY1093884 225mg | BAY1093884 400mg
Number analyzed (Participants) | 8 | 8 | 8
Participants
  TESAEs | 1 | 2 | 1
  Drug-related TESAEs | 0 | 2 | 1

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest
Description: Any thromboembolic or thrombotic microangiopathic event or any hypersensitivity reaction was an adverse event of special interest (AESI). AESIs occurring after the first administration of study drug and up to and including 30 days after the last administration of study drug were defined as treatment-emergent AESIs.
Time Frame: as for outcome 1
Population: Safety analysis set (SAF): all participants with at least one intake of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | BAY1093884 100mg | BAY1093884 225mg | BAY1093884 400mg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 2 | 1

4. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Laboratory Values
Description: "Clinically relevant "implied the presence of a clinical sign or symptom that required medical action.
Time Frame: as for outcome 1
Population: Safety analysis set (SAF): all participants with at least one intake of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | BAY1093884 100mg | BAY1093884 225mg | BAY1093884 400mg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: After the first administration of study drug and up to and including 30 days after the last administration of study drug, with an average of 183 days
Groups:
- BAY1093884 400mg: Subjects received BAY1093884 400 mg once a week until premature termination of the study
Arm/Group | BAY1093884 100mg | BAY1093884 225mg | BAY1093884 400mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/8 | 1/8
Other Adverse Events (participants affected / at risk) | 7/8 | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY1093884 100mg (N=8) | BAY1093884 225mg (N=8) | BAY1093884 400mg (N=8)
Retinal artery thrombosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY1093884 100mg (N=8) | BAY1093884 225mg (N=8) | BAY1093884 400mg (N=8)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 2 (19)
Injection site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 2 (9)
Injection site reaction (General disorders) | 0 (0) | 1 (26) | 0 (0)
Application site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 2 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Acceptable safety and tolerability of befovacimab was not demonstrated in the study, prompting early termination of the study. The "post-hoc" SAP was used for analyses. The other SAP was pre-specified but became not applicable after the termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03597022/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03597022/SAP_001.pdf